CLINICAL TRIAL: NCT04457128
Title: Just-in-Time Adaptive Intervention to Reduce Sedentary Behavior
Brief Title: Real-time Behavioral Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 20-03-3472
Record Dates: First submitted 2020-04-03; First posted 2020-07-07 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-07

CONDITIONS: Cancer; Aging; Comorbidities and Coexisting Conditions
Keywords: physical activity; ecological momentary assessment; health-related quality of life; Just-in-time adaptive intervention
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Micro-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Secular Image (Experimental): Secular Image
  Interventions: Behavioral: Just-in-Time Adaptive Intervention
- Non-secular image (Experimental): non-secular images
  Interventions: Behavioral: Just-in-Time Adaptive Intervention
- Secular message (Experimental): secular messages
  Interventions: Behavioral: Just-in-Time Adaptive Intervention
- Non-secular message (Experimental): non-secular messages
  Interventions: Behavioral: Just-in-Time Adaptive Intervention

INTERVENTIONS:
Behavioral: Just-in-Time Adaptive Intervention — Randomized factorial design

SUMMARY:
The goal of this study is to adapt an evidence-based sedentary behavior reduction intervention for men and women living in Alabama and determine its feasibility, acceptance, and limited efficacy.

DETAILED DESCRIPTION:
The goal of this study is to adapt an evidence-based sedentary behavior reduction intervention for men and women living in Alabama and determine its feasibility, acceptance, and limited efficacy. Community-based Participatory Research methods will be used to adapt an evidence-based curriculum. The adapted curriculum will be delivered via print-based materials and a mobile phone app developed by an external collaborator.

ELIGIBILITY:
Inclusion Criteria:

* • 50 to 75 years old at study enrollment;

  * Currently living in Alabama;
  * Community-dwelling (i.e., not living in an assisted living facility or nursing home);
  * Having access to the internet and a smart phone;
  * Able to perform light-intensity physical activity (i.e., walking);
  * English speaking;
  * Willing to consent to study procedure.

Exclusion Criteria:

* Reporting more than 60 minutes of purposeful physical activity per week;
* Have an unstable mental condition that prevention study activities. Determined by the Physician Health questionnaire.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Usage | 16 weeks
  To percentage of time participants were complying with the study protocol
The Usage, Satisfaction, Ease of use Questionnaire | 16 weeks
  Questionnaire that assesses usage, satisfaction, and ease of use of technology. Each subscale has a maximum score of 20, with higher scores indicating a better outcome.

SECONDARY OUTCOMES:
Change in sedentary time | Week 0 and Week 16
  Accelerometer determined breaks in inactivity during waking hours
Change in light-intensity physical activity | Week 0 and Week 16
  Accelerometer determined activity

CONTACTS AND LOCATIONS:
Overall Officials: Raheem Paxton, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No
No at this time